CLINICAL TRIAL: NCT03325894
Title: A Phase 3, Open-label, Multicenter, 12-Month Safety and Tolerability Study of SHP465 in Children Aged 4 to 12 Years Diagnosed With Attention-deficit/Hyperactivity Disorder
Brief Title: Safety and Tolerability Study of SHP465 in Children Aged 4 to 12 Years Diagnosed With Attention-deficit/Hyperactivity Disorder (ADHD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to efficacy reasons.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP465-308
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD; SHP465; Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SHP465 (Experimental): Group A participants who have been rolled-over from antecedent SHP465 studies and Group B participants who will be newly enrolled into the study will receive SHP465 capsule 6.25 mg orally once daily for 360 days.
  Interventions: Drug: SHP465

INTERVENTIONS:
Drug: SHP465 — SHP465 capsule will be administered in a dose of 6.25 mg orally once daily for 360 days.

SUMMARY:
The purpose of the study is to evaluate the long-term safety and tolerability of SHP465 at 6.25 milligram (mg) in children aged 4 to 12 years diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Participant is male or female aged 4-12 years inclusive at the time of consent.
* Participant's parent or legally authorized representative (LAR) must provide signature of informed consent, and there must be documentation of assent (as applicable) by the participant.
* Participant must meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD (any subtype).
* Participant who is a female and of child-bearing potential must not be pregnant and agree to comply with any applicable contraceptive requirements..
* Participant has an ADHD-RS-5 Child, Home Version Total Score of greater than or equal to (>=) 28 and Clinical Global Impression - Severity of Illness (CGI-S) score >=4 at baseline (Visit 2). Participant is currently not on ADHD therapy, or is not completely satisfied with their current ADHD therapy.

Exclusion Criteria:

* Participant is required or anticipated to take medications that have central nervous system effects or affect performance. Stable use of bronchodilator inhalers is not exclusionary.
* Participant has a concurrent chronic or acute illness, disability, or other condition that might confound the results of safety assessments conducted in the study or that might increase risk to the participant. - Participant has a documented allergy, hypersensitivity, or intolerance to amphetamine or to any excipients in the investigational product.
* Participant has failed to fully respond, based on investigator judgment, to an adequate course of amphetamine therapy.
* Participant has a known family history of sudden cardiac death or ventricular arrhythmia.
* Participant has a blood pressure measurement >=95th percentile for age, sex, and height at screening (Visit 1) and/or baseline (Visit 2).
* Participant has a height less than or equal to (<=) 5th percentile for age and sex at screening (Visit 1) or baseline (Visit 2).
* Participant has a weight <=5th percentile for age and sex at screening (Visit 1) or baseline (Visit 2).
* Participant has a known history of symptomatic cardiovascular disease, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, or other serious cardiac conditions placing them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
* Participant has a history of seizures (other than infantile febrile seizures).
* Participant is taking any medication that is excluded per the protocol.
* Participant had any clinically significant ECG or clinical laboratory abnormalities at the screening (Visit 1) or baseline visit (Visit 2).
* Participant has current abnormal thyroid function, defined as abnormal thyroid-stimulating hormone and thyroxine at the screening or baseline visit. Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
* Participant is currently considered a suicide risk in the opinion of the investigator, has previously made a suicide attempt, or has a prior history of or currently demonstrating suicidal ideation.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2019-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (48):
- United States (48):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - PEWMD, PA, ARCSM, PLLC, PRP, Inc., Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - Riverside Medical Clinic, Riverside, California
  - Peninsula Research Associates - CRN, Rolling Hills, California
  - Pediatric Medical Associates, Sacramento, California
  - Care Research Center, Doral, Florida
  - Power MD Clinical Research Institute, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Acevedo Medical Group, Miami, Florida
  - Pharmacology Research, LLC, Miami, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Clinical Associates of Orlando, Llc, Orlando, Florida
  - GA Psychiatric Services, LLC., Atlanta, Georgia
  - Buford Family Practice, Buford, Georgia
  - One Health Research Clinic, Inc., Norcross, Georgia
  - Institute for Behavioral Medicine, Smyrna, Georgia
  - Advanced Clinical Research, Inc, Meridian, Idaho
  - Conventions Psychiatry and Counseling, Naperville, Illinois
  - Pedia Research, LLC, Evansville, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Qualmedica Research LLC, DBA Pedia Research, Owensboro, Kentucky
  - Neuroscientific Insights, Rockville, Maryland
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - St Charles Psychiatric Associates, Saint Charles, Missouri
  - Alivation Research, LLC., Lincoln, Nebraska
  - Triangle Neuropsychiatry, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - Family Practice Center of Wadsworth, INC., Wadsworth, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Rainbow Research, Inc., Barnwell, South Carolina
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Coastal Pediatric Associates, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Access Clinical Trials, Inc., Nashville, Tennessee
  - El Campo Clinical Trials, El Campo, Texas
  - Houston Clinical Trials, LLC, Houston, Texas
  - Children's Clinic, League City, Texas
  - University of Texas, San Antonio, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - VA South Psychiatric & Family Services, Petersburg, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Mid-Columbia Research, Richland, Washington

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 33 centers in the United States between 02 January 2018 (first participant first visit) and 19 January 2019 (last participant last visit).
Pre-assignment Details: Overall, 141 participants enrolled and received the treatment in two groups (Group A and B). Participants who completed antecedent studies SHP465-112 (NCT03327402) or SHP465-309 (NCT03325881) were in Group A and participants who were directly enrolled into this study were in Group B.
Groups:
- Group A (Antecedent Studies): Participants who completed antecedent studies SHP465-112 (NCT03327402) or SHP465-309 (NCT03325881) were in group A and received 6.25 milligram (mg) SHP465 capsule orally once daily for up to 330 days.
- Group B (Direct Enrollment): Participants who directly enrolled in this study were in group B and received 6.25 mg SHP465 capsule orally once daily for up to 330 days.
Period: Overall Study
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Started | 64 | 77
Completed | 0 | 0
Not Completed | 64 | 77
Not completed — Adverse Event | 2 | 3
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Lost to Follow-up | 4 | 9
Not completed — Lack of Efficacy | 8 | 14
Not completed — Study Terminated by Sponsor | 38 | 43
Not completed — Other (Not received Treatment) | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment) | Total
Number analyzed (Participants) | 63 | 77 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (2.61) | 6.1 (2.33) | 6.8 (2.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 50
  Male | 41 | 49 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 26 | 42
  Not Hispanic or Latino | 46 | 51 | 97
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 17 | 36
  White | 37 | 57 | 94
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs was defined as AEs that start or deteriorate on or after the date of the first dose of investigational product and no later than 3 days following the last dose of investigational product.
Time Frame: From start of study drug administration up to follow-up (approximately up to 367 days)
Population: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
Participants | 29 | 38

2. Primary Outcome: Change From Baseline in Pulse Rate at Final On-Treatment Assessment (FoTA)
Description: Change from baseline in pulse rate at FoTA was reported. FoTA was defined as the last valid assessment obtained after baseline and whilst on investigational product (on or before 2 days after the last dose date). Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product in the current study.
Time Frame: Baseline, FoTA (up to 330 days)
Population: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
beats per minute | 1.5 (9.82) | 0.1 (10.31)

3. Primary Outcome: Change From Baseline in Blood Pressure at Final On-Treatment Assessment (FoTA)
Description: Change from baseline in systolic blood pressure (SBP) and diastolic blood pressure (DBP) at FoTA was reported. FoTA was defined as the last valid assessment obtained after baseline and whilst on investigational product (on or before 2 days after the last dose date). Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product in the current study.
Time Frame: Baseline, FoTA (up to 330 days)
Population: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
Millimeters of mercury
  SBP: Change at FoTA | 0.6 (7.17) | 0.6 (7.36)
  DBP: Change at FoTA | 2.3 (7.76) | 1.7 (6.03)

4. Primary Outcome: Change From Baseline in Height at Final On-Treatment Assessment (FoTA)
Description: Height was measured in centimeters (cm) without shoes and with light clothing using a stadiometer. FoTA was defined as the last valid assessment obtained after baseline and whilst on investigational product (on or before 2 days after the last dose date). Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product in the current study.
Time Frame: Baseline, FoTA (up to 330 days)
Population: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
centimeter | 3.7 (4.60) | 2.9 (2.49)

5. Primary Outcome: Change From Baseline in Weight at Final On-Treatment Assessment (FoTA)
Description: Weight was measured in kilograms (kg) without shoes and with light clothing using a calibrated scale. FoTA was defined as the last valid assessment obtained after baseline and whilst on investigational product (on or before 2 days after the last dose date). Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product in the current study.
Time Frame: Baseline, FoTA (up to 330 days)
Population: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
kilograms | 1.4 (2.93) | 1.1 (2.41)

6. Primary Outcome: Change From Baseline in Hematology Parameters at Early Termination/Day 360
Description: Change from baseline in hematology parameter basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils band form, segmented neutrophils, neutrophils/total cells and platelets were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study. Here, the number of participants analyzed refer to the participants evaluable for this outcome at specific categories.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
10^9 cells per liter
  Basophils: number analyzed (Participants) | 30 | 31
  Basophils | -0.01 (0.040) | 0.01 (0.051)
  Eosinophils: number analyzed (Participants) | 30 | 31
  Eosinophils | 0.02 (0.389) | 0.04 (0.240)
  Leukocytes: number analyzed (Participants) | 31 | 31
  Leukocytes | -0.25 (1.519) | -0.09 (2.107)
  Lymphocytes: number analyzed (Participants) | 30 | 31
  Lymphocytes | 0.14 (0.948) | -0.12 (0.685)
  Monocytes: number analyzed (Participants) | 30 | 31
  Monocytes | -0.12 (0.282) | 0.01 (0.217)
  Neutrophils Band Form: number analyzed (Participants) | 15 | 22
  Neutrophils Band Form | 0.00 (0.00) | 0.00 (0.049)
  Segmented Neutrophils: number analyzed (Participants) | 15 | 22
  Segmented Neutrophils | -0.40 (1.296) | -0.02 (2.139)
  Neutrophils/Total Cells: number analyzed (Participants) | 31 | 31
  Neutrophils/Total Cells | -0.32 (1.349) | 0.00 (1.915)
  Platelets: number analyzed (Participants) | 29 | 31
  Platelets | 8.0 (46.76) | 4.6 (60.19)

7. Primary Outcome: Change From Baseline in Leukocytes at Early Termination/Day 360
Description: Change from baseline in hematology leukocytes parameter: basophils, eosinophils, lymphocytes, monocytes and neutrophil were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of leukocytes
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
percentage of leukocytes
  Basophils/Leukocytes: number analyzed (Participants) | 31 | 31
  Basophils/Leukocytes | -0.17 (0.631) | 0.04 (0.589)
  Eosinophils/Leukocytes: number analyzed (Participants) | 31 | 31
  Eosinophils/Leukocytes | 0.38 (4.288) | 0.30 (3.222)
  Lymphocytes/Leukocytes: number analyzed (Participants) | 31 | 31
  Lymphocytes/Leukocytes | 4.42 (12.140) | -0.97 (11.517)
  Monocytes/Leukocytes: number analyzed (Participants) | 31 | 31
  Monocytes/Leukocytes | -1.02 (3.982) | 0.52 (2.650)
  Neutrophils Band Form/Leukocytes: number analyzed (Participants) | 16 | 22
  Neutrophils Band Form/Leukocytes | 0.0 (0.00) | 0.0 (0.62)
  Neutrophils, Segmented/Leukocytes: number analyzed (Participants) | 16 | 22
  Neutrophils, Segmented/Leukocytes | -3.8 (12.39) | -0.6 (13.15)
  Neutrophils/Leukocytes: number analyzed (Participants) | 31 | 31
  Neutrophils/Leukocytes | -3.62 (13.359) | 0.35 (11.756)

8. Primary Outcome: Change From Baseline in Erythrocytes at Early Termination/Day 360
Description: Change from baseline in hematology parameter erythrocytes were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study. Here, the number of participants analyzed refer to the participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 31 | 31
10^12 cells per liter | 0.017 (0.3368) | -0.007 (0.2889)

9. Primary Outcome: Change From Baseline in Erythrocytes Mean Corpuscular Hemoglobin Concentration at Early Termination/Day 360
Description: Change from baseline in hematology parameter erythrocytes mean corpuscular hemoglobin concentration were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study.Here, the number of participants analyzed refer to the participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Deviation); unit: gram per deciliter
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 31 | 31
gram per deciliter | -0.09 (0.664) | -0.16 (1.018)

10. Primary Outcome: Change From Baseline in Erythrocytes Mean Corpuscular Hemoglobin at Early Termination/Day 360
Description: Change from baseline in hematology parameter erythrocytes mean corpuscular hemoglobin were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: picogram
Groups:
- Group A (Antecedent Studies): Participants in group A received 6.25 milligram (mg) SHP465 capsule orally once daily for up to 330 days.
- Group B (Direct Enrollment): Participants in group B received 6.25 mg SHP465 capsule orally once daily for up to 330 days.
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 31 | 31
picogram | 0.42 (0.642) | 0.38 (1.259)

11. Primary Outcome: Change From Baseline in Hematocrit at Early Termination/Day 360
Description: Change from baseline in hematology parameter hematocrit were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage of hematocrit
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 31 | 31
percentage of hematocrit | 0.86 (2.784) | 0.59 (2.901)

12. Primary Outcome: Change From Baseline in Hemoglobin at Early Termination/Day 360
Description: Change from baseline in hematology parameter hemoglobin were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 31 | 31
gram per liter | 2.5 (8.68) | 1.5 (9.82)

13. Primary Outcome: Change From Baseline in Hematology Parameters (Erythrocytes Mean Corpuscular Volume and Mean Platelet Volume) at Early Termination/ Day 360
Description: Change from baseline in hematology parameter erythrocytes mean corpuscular volume and mean platelet volume were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
femtoliters
  Erythrocytes Mean Corpuscular Volume: number analyzed (Participants) | 31 | 31
  Erythrocytes Mean Corpuscular Volume | 1.48 (1.438) | 1.46 (2.565)
  Mean Platelet Volume: number analyzed (Participants) | 29 | 31
  Mean Platelet Volume | -0.1 (0.77) | 0.2 (0.96)

14. Primary Outcome: Change From Baseline in Chemistry Parameters at Early Termination/Day 360
Description: Change from baseline in chemistry parameter alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, gamma glutamyl transferase, and lactate dehydrogenase were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Unit per liter
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
Unit per liter
  Alanine Aminotransferase: number analyzed (Participants) | 32 | 30
  Alanine Aminotransferase | -2.3 (4.18) | 9.6 (52.75)
  Alkaline Phosphatase: number analyzed (Participants) | 32 | 30
  Alkaline Phosphatase | -18.2 (62.28) | -32.6 (68.15)
  Aspartate Aminotransferase: number analyzed (Participants) | 32 | 30
  Aspartate Aminotransferase | -1.9 (5.27) | 21.4 (129.48)
  Gamma Glutamyl Transferase: number analyzed (Participants) | 32 | 30
  Gamma Glutamyl Transferase | -0.4 (2.20) | 1.3 (5.06)
  Lactate Dehydrogenase: number analyzed (Participants) | 22 | 30
  Lactate Dehydrogenase | -9.0 (24.24) | 26.2 (185.52)

15. Primary Outcome: Change From Baseline in Chemistry Parameters (Albumin and Protein) at Early Termination/Day 360
Description: Change from baseline in chemistry parameters albumin and protein were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: gram per liter
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 32 | 30
gram per liter
  Albumin | -0.2 (2.82) | -0.1 (2.45)
  Protein | 0.7 (4.27) | 1.0 (3.55)

16. Primary Outcome: Change From Baseline in Chemistry Parameters (Blood Urea Nitrogen, Cholesterol, Glucose, Phosphate, Potassium, Sodium and Urate) at Early Termination/Day 360
Description: Change from baseline in chemistry parameters blood urea nitrogen, cholesterol, glucose, phosphate, potassium, sodium and urate were studies. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
millimoles per liter
  Blood Urea Nitrogen: number analyzed (Participants) | 32 | 30
  Blood Urea Nitrogen | -0.235 (1.0664) | -0.036 (1.4248)
  Calcium: number analyzed (Participants) | 31 | 30
  Calcium | 0.035 (0.1101) | 0.004 (0.0977)
  Cholesterol: number analyzed (Participants) | 23 | 30
  Cholesterol | -0.082 (0.4592) | -0.295 (0.8294)
  Glucose: number analyzed (Participants) | 32 | 30
  Glucose | -0.183 (0.9841) | 0.138 (0.9205)
  Phosphate: number analyzed (Participants) | 31 | 30
  Phosphate | -0.045 (0.1940) | -0.153 (0.2056)
  Potassium: number analyzed (Participants) | 31 | 30
  Potassium | -0.02 (0.569) | -0.01 (0.367)
  Sodium: number analyzed (Participants) | 32 | 30
  Sodium | 0.8 (2.57) | 0.3 (2.48)
  Urate: number analyzed (Participants) | 32 | 30
  Urate | -0.0073 (0.04488) | 0.0142 (0.07180)

17. Primary Outcome: Change From Baseline in Chemistry Parameters (Bilirubin and Creatinine) at Early Termination/Day 360
Description: Change from baseline in chemistry parameters bilirubin and creatinine were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: micromoles per liter
Groups:
- Group A (Antecedent Study): Participants who completed antecedent studies SHP465-112 (NCT03327402) or SHP465-309 (NCT03325881) were in group A and received 6.25 milligram (mg) SHP465 capsule orally once daily for up to 330 days.
Arm/Group | Group A (Antecedent Study) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
micromoles per liter
  Bilirubin: number analyzed (Participants) | 27 | 25
  Bilirubin | 0.90 (3.644) | -0.14 (2.994)
  Creatinine: number analyzed (Participants) | 32 | 29
  Creatinine | 3.3 (8.20) | 6.7 (17.15)

18. Primary Outcome: Change From Baseline in Thyrotropin at Early Termination/ Day 360
Description: Change from baseline in thyrotropin were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milli-international units per litre
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 30 | 25
milli-international units per litre | 0.2576 (0.98862) | 0.2392 (0.90169)

19. Primary Outcome: Change From Baseline in Thyroxine,Free at Early Termination/Day 360
Description: Change from baseline in thyroxine,free were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: picomole per liter
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 21 | 25
picomole per liter | 0.61 (1.851) | -0.46 (2.632)

20. Primary Outcome: Change From Baseline in Urinalysis (Specific Gravity) at Early Termination/Day 360
Description: Change from baseline in urine specific gravity were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 30 | 35
Ratio | 0.0029 (0.00762) | 0.0010 (0.00923)

21. Primary Outcome: Change From Baseline in Urobilinogen at Early Termination/Day 360
Description: Change from baseline in urobilinogen were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early termination/Day 360
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 21 | 34
milligrams per deciliter | 0.09 (0.393) | 0.05 (0.309)

22. Primary Outcome: Change From Baseline in Urine Potential of Hydrogen (pH) at Early Termination/Day 360
Description: Change from baseline in urine pH were reported. Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: Baseline, Early Termination/Day 360
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 30 | 35
pH | 0.1 (0.83) | 0.1 (1.07)

23. Primary Outcome: Change From Baseline in Heart Rate at Final On-Treatment Assessment (FoTA)
Description: Heart rate was measured by Electrocardiogram (ECG). ECG was performed using the central ECG provider's equipment and was send to the central ECG provider electronically. Change from baseline in heart rate at FoTA were reported. FoTA was defined as the last valid assessment obtained after baseline and whilst on investigational product (on or before 2 days after the last dose date). Group A baseline was the baseline of the antecedent studies. Group B baseline was the average of all valid ECG measurements as the last assessment obtained before the first dose of investigational product.
Time Frame: Baseline, FoTA (up to 330 days)
Population: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 61 | 75
beats per minute | 1.78 (7.618) | -0.12 (10.973)

24. Primary Outcome: Change From Baseline in Electrocardiogram Parameters at Final On-Treatment Assessment (FoTA)
Description: ECG was performed using the central ECG provider's equipment and was sent to the central ECG provider electronically to measure PR, RR, QRS , QT, QTcB and QTcF intervals. FoTA was defined as the last valid assessment obtained after Baseline and whilst on investigational product (on or before 2 days after the last dose date).Group A baseline was the baseline of the antecedent studies. Group B baseline was the average of all valid ECG measurements as the last assessment obtained before the first dose of investigational product.
Time Frame: Baseline, FoTA (up to 330 days)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 61 | 75
milliseconds
  FoTA: PR Interval | -1.77 (10.129) | 0.14 (8.539)
  FoTA: RR Interval | -18.05 (71.382) | -1.77 (88.658)
  FoTA: QRS Interval | 0.93 (4.419) | 1.62 (5.688)
  FoTA: QT Interval | -4.74 (17.826) | -1.49 (18.616)
  FoTA: QTcB Interval | -0.52 (14.145) | -1.39 (14.796)
  FoTA: QTcF Interval | -1.97 (13.126) | -1.37 (11.808)

25. Primary Outcome: Number of Participants With Quality of Sleep Assessed by Post Sleep Questionnaire (PSQ) at Final On-Treatment Assessment (FoTA)
Description: PSQ was a 7-item questionnaire typically used to assess sleep quality with pharmacologic treatment. The questionnaire collects data on average time to sleep, sleep latency, frequency of interrupted sleep, duration of interrupted sleep, total sleep time and sleep quality over the last week. The assessment was done by the nature of the responses, not by a numbered scale. Participants analyzed for number of times woke up per night category were only the participants who responded as yes for the woke up during the night category in this outcome measure. FoTA was defined as the last valid assessment obtained after Baseline and whilst on investigational product (on or before 2 days after the last dose date). Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product.
Time Frame: FoTA (up to 330 days)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
Participants
  FoTA: Woke up during the night - Yes | 17 | 13
  FoTA: Woke up during the night - No | 46 | 64
  FoTA: Number of times woke up per night = 0: number analyzed (Participants) | 17 | 14
  FoTA: Number of times woke up per night = 0 | 0 | 2
  FoTA: Number of times woke up per night = 1: number analyzed (Participants) | 17 | 14
  FoTA: Number of times woke up per night = 1 | 12 | 10
  FoTA: Number of times woke up per night = 2: number analyzed (Participants) | 17 | 14
  FoTA: Number of times woke up per night = 2 | 4 | 2
  FoTA: Number of times woke up per night = 3: number analyzed (Participants) | 17 | 14
  FoTA: Number of times woke up per night = 3 | 1 | 0
  FoTA: Number of times woke up per night = 4: number analyzed (Participants) | 17 | 14
  FoTA: Number of times woke up per night = 4 | 0 | 0
  FoTA: Number of times woke up per night >= 5: number analyzed (Participants) | 17 | 14
  FoTA: Number of times woke up per night >= 5 | 0 | 0
  FoTA: Overall quality of sleep - Very Poor | 0 | 0
  FoTA: Overall quality of sleep - Poor | 6 | 1
  FoTA: Overall quality of sleep - Average | 23 | 20
  FoTA: Overall quality of sleep - Good | 24 | 29
  FoTA: Overall quality of sleep - Very Good | 10 | 27
  FoTA: Past week a typical week - Yes | 48 | 66
  FoTA: Past week a typical week - No | 15 | 11
  FoTA: Past week was not typical - Vacation: number analyzed (Participants) | 15 | 11
  FoTA: Past week was not typical - Vacation | 4 | 1
  FoTA: Past week was not typical - School break: number analyzed (Participants) | 15 | 11
  FoTA: Past week was not typical - School break | 7 | 7
  FoTA: Past week was not typical - Friend house: number analyzed (Participants) | 15 | 11
  FoTA: Past week was not typical - Friend house | 0 | 0
  FoTA: Past week was not typical - ill: number analyzed (Participants) | 15 | 11
  FoTA: Past week was not typical - ill | 0 | 2
  FoTA: Past week was not typical - other: number analyzed (Participants) | 15 | 11
  FoTA: Past week was not typical - other | 4 | 1
  FoTA: Overall quality - Better than usual: number analyzed (Participants) | 19 | 12
  FoTA: Overall quality - Better than usual | 1 | 0
  FoTA: Overall quality - Same as usual: number analyzed (Participants) | 19 | 12
  FoTA: Overall quality - Same as usual | 13 | 8
  FoTA: Overall quality - Worse than usual: number analyzed (Participants) | 19 | 12
  FoTA: Overall quality - Worse than usual | 5 | 4

26. Primary Outcome: Length of Time Awake Per Night and Length of Time to Fall Asleep Per Night Assessed by Post Sleep Questionnaire (PSQ) at Final On-Treatment Assessment (FoTA)
Description: PSQ was a 7-item questionnaire typically used to assess sleep quality with pharmacologic treatment. The questionnaire collects data on average time to sleep, sleep latency, frequency of interrupted sleep, duration of interrupted sleep, total sleep time and sleep quality over the last week. FoTA was defined as the last valid assessment obtained after Baseline and whilst on investigational product (on or before 2 days after the last dose date). Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product. Length of time awake per night and length of time to fall asleep per night was assessed at FoTA.
Time Frame: FoTA (up to 330 days)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
minutes
  Length of Time to Fall Asleep per Night | 20.2 (17.12) | 22.3 (24.74)
  Length of Time Awake per Night: number analyzed (Participants) | 17 | 14
  Length of Time Awake per Night | 8.8 (4.14) | 14.4 (23.10)

27. Primary Outcome: Length of Time Sleeping Per Night Assessed by Post Sleep Questionnaire (PSQ) at Final On-Treatment Assessment (FoTA)
Description: PSQ was a 7-item questionnaire typically used to assess sleep quality with pharmacologic treatment. The questionnaire collects data on average time to sleep, sleep latency, frequency of interrupted sleep, duration of interrupted sleep, total sleep time and sleep quality over the last week. FoTA was defined as the last valid assessment obtained after Baseline and whilst on investigational product (on or before 2 days after the last dose date). Group A baseline was the baseline of the antecedent studies. Group B baseline was the last value collected before the first dose of investigational product. Length of time sleeping per night was assessed at FoTA.
Time Frame: FoTA (up to 330 days)
Population: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 63 | 77
hours | 9.1 (1.40) | 9.6 (1.21)

28. Primary Outcome: Total Sleep Disturbance Score of Children's Sleep Habits Questionnaire (CSHQ ) at Final On-Treatment Assessment (FoTA)
Description: CSHQ was a tool designed to screen for the most common sleep problems in children and consisted of 33 items for scoring and several extra items intended to provide administrators with other potentially useful information about respondents. The instrument evaluates the 8 different subscales: bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep disordered breathing, and daytime sleepiness. A 3-point scale was used for rating: "usually" if the sleep behavior occurs 5 to 7 times per week, "sometimes" for 2 to 4 times per week, and "rarely" for once or not at all during the week. The TSD score, which is the sum of all responses, included all items of the 8 subscales, but consisted of only 33 items because two on the bedtime resistance and sleep anxiety subscales were identical (range: 0, 99). A negative value indicates less sleep disturbance.
Time Frame: FoTA (up to 330 days)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 62 | 77
Units on scale | 42.2 (8.44) | 39.3 (5.85)

29. Primary Outcome: Number of Participants With a Positive Response in Columbia-Suicide Severity Rating Scale (C-SSRS) at Day 330
Description: C-SSRS is a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The number of participants with postive response in suicidal ideation and suicidal behavior were reported.
Time Frame: Day 330
Population: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study.. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 2 | 2
Participants
  Suicidal Ideation: number analyzed (Participants) | 0 | 0
  Suicidal Ideation | 0 | 0
  Suicidal Behavior | 0 | 0

30. Secondary Outcome: Change From Baseline in Clinician-administered Attention-Deficit/Hyperactivity Disorder Rating Scale-5 (ADHD-RS-5) Total Score at Final On-Treatment Assessment (FoTA)
Description: Clinician administered ADHD-RS-5, child, home version total score were analyzed. ADHD-RS-5 consists of 18 items designed to reflect current symptomatology of ADHD based on diagnostic and statistical manual of mental disorders, fifth edition (DSM-5) criteria. Each item is scored on a 4-point scale ranging from 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54. The 18 items may be grouped into 2 subscales: hyperactivity/impulsivity (9 items) and inattentiveness (9 items). Higher total scores indicated higher impairment and lower scores indicated no impairment. FoTA was defined as the last valid assessment obtained after Baseline and whilst on investigational product (on or before 2 days after the last dose date).
Time Frame: Baseline, FoTA (up to 330 days)
Population: Full analysis set (FAS) consisted of all participants in the safety set who have completed at least 1 post-dose efficacy assessment using ADHD-RS-5 Total Score. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 62 | 77
Score on a scale | -19.2 (1.88) | -19.3 (1.69)

31. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) at Final On-Treatment Assessment (FoTA)
Description: CGI-I scale was performed to rate the improvement of a participant's condition on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). FoTA was defined as the last valid assessment obtained after baseline and whilst on investigational product (on or before 2 days after the last dose date).
Time Frame: FoTA (up to 330 days)
Population: FAS consisted of all participants in the safety set who have completed at least 1 post-dose efficacy assessment using ADHD-RS-5 Total Score. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
Number analyzed (Participants) | 62 | 77
Score on a scale | 2.7 (0.16) | 2.9 (0.15)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (approximately up to 367 days)
Description: Safety set consisted of all participants who had taken at least 1 dose of investigational product in this current study.
Arm/Group | Group A (Antecedent Studies) | Group B (Direct Enrollment)
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/63 | 1/77
Other Adverse Events (participants affected / at risk) | 12/63 | 20/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Antecedent Studies) (N=63) | Group B (Direct Enrollment) (N=77)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Antecedent Studies) (N=63) | Group B (Direct Enrollment) (N=77)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 7 (12)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (5)
Weight decreased (Investigations) | 3 (4) | 6 (7)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 6 (7)
Headache (Nervous system disorders) | 5 (5) | 3 (4)
Irritability (Psychiatric disorders) | 4 (5) | 1 (1)

LIMITATIONS AND CAVEATS:
The FDA agreed that this 12-month, open-label, long-term safety study (SHP465-308) should be terminated early due to the lack of efficacy observed in the 4-week efficacy and safety study SHP465-309 (NCT03325881).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT03325894/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT03325894/SAP_001.pdf